CLINICAL TRIAL: NCT02678533
Title: Pilot Study Assessing the Feasibility of CD34+ Cells Mobilization and Collection After Treatment With G-CSF and Plerixafor in Patients With Fanconi Anemia for Subsequent Treatment by Gene Therapy
Brief Title: Mobilization and Collection of Peripheral Blood Stem Cells in Patients With Fanconi Anemia Using G-CSF and Plerixafor
Acronym: FancoMob
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: EuroFancolen (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130103; 2014-005264-14 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Fanconi Anemia
Keywords: Fanconi Anemia; CD34+ cells mobilization; G-CSF; Plerixafor; gene therapy
MeSH Terms: conditions — Fanconi Anemia | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fanconi anemia (Experimental): G-CSF and Plerixafor
  Interventions: Drug: G-CSF; Drug: Plerixafor

INTERVENTIONS:
Drug: G-CSF — D1 to D4 : Injection of 12 µg/kg of G-CSF twice a day . D5 : injection of 12 µg/kg of G-CSF (once/ twice a day according to cytapheresis's realization)
Drug: Plerixafor — D5 : injection of 24mg/kg of plerixafor once a day until cytapheresis has be done (maximum of 4 days)

SUMMARY:
The purpose of this study is to assess the feasibility of Plerixafor used in combination with G-CSF (Granulocyte Colony Stimulating Factor) in 5 Fanconi anemia patients to mobilize and collect a sufficient number of peripheral blood CD34+ cells for peripheral blood apheresis, for further gene therapy study.

DETAILED DESCRIPTION:
Fanconi anemia is an autosomal recessive disease with an average survival of around 24 years old. The number of cells producted by bone marrow decreases around 5-10 years old. Hematological symptoms occur around 7 years old. 80% of patients with Fanconi anemia have clinical signs of bone marrow failure in the first decade of life. Generally macrocytosis is the first noticeable sign. Then it leads to thrombocytopenia, anemia and pancytopenia.

Epidemiologic studies show that nearly all of the patients will have medullar aplasia before 40 years old, which is then the first cause of mortality.

It must be emphasized that these complications may occur simultaneously for the same patient, so joint therapeutic intervention is needed.

There is no basic treatment. Some currently used treatments cure cytopenias. These treatments involve blood transfusion, oral androgen, hematopoietic growth factor administration, such as Epo and G-CSF to treat anemia and neutropenia. These treatments are not curative. Hematopoietic stem cell transplantation is the only treatment able to restore permanently hematopoiesis. However, this treatment leads to a high level risk of developing solid tumors and other complications.

All these data justify of developing a stem cells gene therapy treatment using a lentiviral vector expressing wild-type FANCA gene under CIBER promoter.

Three studies have shown the potential number of cells to be mobilized in patients with Fanconi anemia.

The aim is first, to show if administering G-CSF with plerixafor may lead to collect enough cells to potentially perform a gene therapy graft. Secondly the study will assess the tolerance, the stem cells' mobilization kinetic and collected cells' biological features.

This study will be performed in Necker Children Hospital. 8 patients will be enrolled in order to reach 5 treated patients and to analyse how many injections and days are required to reach the cells' number goal.

Sequential blood samples of patients will be drawn to monitor complete blood count (CBC), platelet, CD34+ cells rate and stem cells phenotype.

The clinical and biological data will be anonymously entered in a electronic case report by the investigators up to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Fanconi anemia
* Patient from 2 to 17 years old
* Potential indication for allogenic bone arrow graft without HLA-identical brotherhood available
* Patient's weight >10kg
* Treated and followed for at least the previous two years in a specialized center where they got a full assessment of their disease
* For women of childbearing age, not pregnant and use of an effective contraception during the entire participation in the research.
* Affiliated or beneficiary of an health insurance regimen
* Informed and signed consent

Exclusion Criteria:

* Patient unable to follow the visits required by the protocol
* Positive serology for HIV-1/2, HTLV-1/2, HCV and HbS
* Bacterial, viral, fungal or parasitic active infection with clinical signs
* Personal history of cancer, myeloproliferative hematopathy or immune deficiency
* Heart failure and / or heart rhythm disorder
* History of allogeneic graft of hematopoietic stem cells
* Patient with an HLA-identical brotherhood donor available
* Myelodysplasia diagnose on myelogram
* Cytogenetic abnormality on karyotype
* Malignant solid tumor
* Documented spontaneous genetic reversion of medullary process
* Diagnosis of a psychiatric disorder that could compromise his/her ability to participate in the study
* Any disorder according to the investigator, that could compromise the ability of patient to give his writing consent and/or to comply with requiring study's procedures
* Current Pregnancy
* Heart, kidney or liver failure
* Current participation in another interventional clinical trial
* Patient under Medical Assistance State
* Hypersensitivity to plerixafor or any excipient contained in MOZOBIL®
* Hypersensitivity to filgrastim or any of its' excipient

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
level of CD34+ cells mobilization | from day 5 to day 8 after the first injection of G-CSF

SECONDARY OUTCOMES:
number of treatment-related adverse events as a measure of tolerability | 30 days after cytapheresis
  Occurrence of adverse effect due to G-CSF and plerixafor administration

CONTACTS AND LOCATIONS:
Overall Officials: Marina CAVAZZANA, MD, PhD, Study Director — AP-HP, Necker hospital
Locations (1):
- Hôpital necker-Enfants malades, Paris, PARIS, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diana JS, Manceau S, Leblanc T, Magnani A, Magrin E, Bendavid M, Couzin C, Joseph L, Soulier J, Cavazzana M, Lefrere F. A new step in understanding stem cell mobilization in patients with Fanconi anemia: A bridge to gene therapy. Transfusion. 2022 Jan;62(1):165-172. doi: 10.1111/trf.16721. Epub 2021 Nov 9. PMID 34751952